CLINICAL TRIAL: NCT04940481
Title: TROLLEY Study - TRansit Opportunities for HeaLth, Livability, Exercise and EquitY
Acronym: TROLLEY
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Katie Crist, Assistant Project Scientist, University of California, San Diego
Other Study IDs: 78646
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Physical Activity
Keywords: active travel, equity, commute mode
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The researchers are evaluating longitudinal changes in multiple health, economic, and environmental outcomes over a 3-year COVID recovery period and in the context of a new light rail transit (LRT) line, called the Mid-Coast Trolley, among 465 UC San Diego (UCSD) staff. The primary aim is to evaluate change in objectively measured total and moderate to vigorous physical activity (MVPA), travel mode, and vehicle miles traveled (VMT).

ELIGIBILITY:
Inclusion Criteria:

1. are 18 years of age or older;
2. are a full or part-time employee at UC San Diego
3. Prior to COVID-19, you used to commute to La Jolla at least 2 days per week;
4. have lived in the neighborhood selected for the study for at least one year;
5. are able to walk without human assistance;
6. are comfortable reading and writing in English or Spanish;
7. have a reliable phone where you can be reached;
8. spend most of your time in San Diego County;
9. don't plan on moving in the next year;
10. are able to give informed consent and comply with the protocol;
11. are willing to complete all assessments and wear all devices for 7 days at 3 different time points in the next 2 years.

Exclusion Criteria:

1) pregnant, 2) mental state that would preclude understanding the protocol, 3) medical condition that would affect physical activity, 4) taking part in another physical activity related research study, and 5) live or regularly travel outside of San Diego County.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will study UCSD staff. We will aim to recruit 50% from people of color, and 50% low income (<80% Area Median Income), 50% female, and 50% living within 1 mile of a transit stop that connects to the Mid-Coast Trolley.
Sampling Method: Non-Probability Sample
Enrollment: 479 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2025-06-14 (Estimated); Study Completion 2025-06-14 (Estimated)

PRIMARY OUTCOMES:
Moderate to vigorous physical activity | 2 years
  Minutes

SECONDARY OUTCOMES:
Active commute mode | 2 years
  %

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego, La Jolla, California, United States

REFERENCES:
- [Background] Crist K, Benmarhnia T, Frank LD, Song D, Zunshine E, Sallis JF. The TROLLEY Study: assessing travel, health, and equity impacts of a new light rail transit investment during the COVID-19 pandemic. BMC Public Health. 2022 Aug 2;22(1):1475. doi: 10.1186/s12889-022-13834-1. PMID 35918683
- See also: TROLLEY study protocol paper — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9344230/